CLINICAL TRIAL: NCT04166630
Title: Accelerometer Motion to Measure Muscle Fatigue in Critically Ill Patients
Brief Title: Diagnosing Intensive Care Unit (ICU) Acquired Weakness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Randi Smith, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00109793
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Results first posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-07

CONDITIONS: ICU Acquired Weakness
Keywords: Biofeedback; Muscular disorders; Neuromuscular disorders; Rehabilitation
MeSH Terms: conditions — Muscular Diseases; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ICU Acquired Weakness Group (Experimental): Participants with a score less than 48 on the Medical Research Council (MRC) Scale will be classified as having ICU acquired weakness. All participants will have their skeletal muscles tested with a clinical electrical stimulator.
  Interventions: Device: Clinical Electrical Stimulator
- No ICU Acquired Weakness Group (Experimental): Participants with a score of 48 or greater on the Medical Research Council (MRC) Scale will be classified as not having ICU acquired weakness. All participants will have their skeletal muscles tested with a clinical electrical stimulator.
  Interventions: Device: Clinical Electrical Stimulator

INTERVENTIONS:
Device: Clinical Electrical Stimulator — Conductive electrodes will be on the skin at each end of the tested muscle(s). Each subject will have two target muscle groups tested (extensor carpi radialis longus, and tibialis anterior). Each muscle will be stimulated at three separate stimulation frequencies (2 Hz, 4 Hz, and 6Hz) over 3 minutes each, for a total of 9 minutes of stimulation per muscle. The clinical electrical stimulator will deliver mild electrical stimulations to the muscle (20-100 mA).
  Other Names: Vectra Genisys Therapy System

SUMMARY:
The goal of this study is to develop a non-invasive test to diagnose intensive care unit (ICU) acquired weakness that can be administered to both responsive and non-responsive patients. Study participation will involve the measurement of muscle fatigue during a single 30 minute session. Skeletal muscle will be stimulated with an FDA approved clinical electrical stimulator and accelerations will be passively recorded with an accelerometer.

DETAILED DESCRIPTION:
The primary purpose of this study is to develop a procedure to identify intensive care unit (ICU) acquired weakness. This condition occurs in a subset of people admitted into the ICU, and is associated with a 30% increased risk of death before discharge from the ICU. There are currently major limitations in the ability to diagnose ICU acquired weakness, making it difficult to study. The goal is to develop a non-invasive test that can be administered to both responsive and non-responsive patients. The current proposal will focus on replicating the results of previous research using motion detecting accelerometers to measure fatigue in human skeletal muscles. This study is designed to test out the procedures in patients who have been transferred from the ICU to a lower level of care so that follow-on studies can be designed to help mitigate this condition in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients transferred from the ICU to a lower level of care within the past 7 days
* Mechanical ventilation for greater than 7 days while in the ICU
* Ability to understand English and provide written consent

Exclusion Criteria:

* Vulnerable populations including: patients who are pregnant or prisoners
* Patients who are unable to understand English or provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randi Smith, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the publications will be available for sharing, after deidentification.
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing beginning 9 months after article publication and ending 36 months following article publication.
Access Criteria: Data will be available for sharing with investigators whose proposed used of the data has been approved for meta-analysis. Information regarding submitting proposals and accessing data will be available by contacting the study staff (contact information to be provided).

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ICU Acquired Weakness Group | No ICU Acquired Weakness Group
Started | 5 | 17
Completed | 5 | 16
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ICU Acquired Weakness Group | No ICU Acquired Weakness Group | Total
Number analyzed (Participants) | 5 | 17 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 14 | 17
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (21.3) | 44.6 (21.4) | 45.5 (21.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 15 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 5 | 13 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 11 | 16
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 17 | 22

OUTCOME MEASURES:

1. Primary Outcome: Peak Acceleration Measured in Extensor Carpi Radialis Longus
Description: The highest acceleration over a single muscle twitch will be used as the peak acceleration. Peak acceleration will be measured in acceleration in number of times gravity (g). Higher twitch acceleration is a better response.
Time Frame: Day 1
Population: 2 subjects data sets in the No ICU Acquired Weakness Group, were lost due to device malfunction. One additional subject had no data due to a malfunction with the accelerometer firmware The device manufacturer was contacted and were able to update the device, but no data was recorded during that trial.
Measure: Mean (Standard Deviation); unit: units of Gravity
Arm/Group | ICU Acquired Weakness Group | No ICU Acquired Weakness Group
Number analyzed (Participants) | 5 | 13
units of Gravity
  Twitch acceleration at 20 Hz | 0.476 (0.467) | 1.639 (0.772)
  Twitch acceleration at 40 Hz | 0.541 (0.591) | 1.608 (0.803)
  Twitch acceleration at 60Hz | 0.373 (0.402) | 1.300 (0.662)

2. Primary Outcome: Peak Acceleration Measured in Tibialis Anterior
Description: as for outcome 1
Time Frame: Day 1
Population: 1 subject data set in the No ICU Acquired Weakness Group, could not be analyzed due to excessive subject motion during the trial. One additional subject had no data due to a malfunction with the accelerometer firmware The device manufacturer was contacted and were able to update the device, but no data was recorded during that trial.
Measure: Mean (Standard Deviation); unit: Units of Gravity
Arm/Group | ICU Acquired Weakness Group | No ICU Acquired Weakness Group
Number analyzed (Participants) | 5 | 14
Units of Gravity
  Twitch acceleration at 20 Hz | 0.105 (0.151) | 1.115 (0.677)
  Twitch acceleration at 40 Hz | 0.102 (0.144) | 1.029 (0.585)
  Twitch acceleration at 60 Hz | 0.101 (0.153) | 0.593 (0.494)

3. Primary Outcome: Time to Peak Acceleration Measured in Extensor Carpi Radialis Longus
Description: The time, in seconds, until peak acceleration is reached will be assessed at 2, 4 and 6 Hz. There is not a reference range for the time to peak force and at this time it is unclear if a shorter or longer time to peak force indicates a more desirable state of health.
Time Frame: Day 1 at 2 Hz, Day 1 at 4 Hz, Day 1 at 6 Hz
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | ICU Acquired Weakness Group | No ICU Acquired Weakness Group
Number analyzed (Participants) | 5 | 13
Seconds
  Day 1 at 2 Hz | 64.7 (69.3) | 119.5 (55.1)
  Day 1 at 4 Hz | 9.8 (14.1) | 64.6 (56.2)
  Day 1 at 6 Hz | 1.5 (1.8) | 33.7 (53.2)

4. Primary Outcome: Time to Peak Acceleration Measured in Tibialis Anterior
Description: The time, in seconds, until peak acceleration is reached will be assessed. There is not a reference range for the time to peak force and at this time it is unclear if a shorter or longer time to peak force indicates a more desirable state of health.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | ICU Acquired Weakness Group | No ICU Acquired Weakness Group
Number analyzed (Participants) | 5 | 14
Seconds
  Day 1 at 2 Hz | 45.5 (68.6) | 100.1 (53.0)
  Day 1 at 4 Hz | 22.0 (47.9) | 32.3 (43.3)
  Day 1 at 6 Hz | 8.8 (19.6) | 19.3 (27.1)

5. Primary Outcome: End Acceleration Measured in Extensor Carpi Radialis Longus
Description: End acceleration is the twitch acceleration averaged over 5 twitches over the last second of stable twitches within the stimulation period. A reference range has not yet been established for this measurement.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units of Gravity
Arm/Group | ICU Acquired Weakness Group | No ICU Acquired Weakness Group
Number analyzed (Participants) | 5 | 13
Units of Gravity
  Twitch acceleration at 20 Hz | 0.289 (0.328) | 1.383 (0.524)
  Twitch acceleration at 40 Hz | 0.147 (0.161) | 1.021 (0.755)
  Twitch acceleration at 60 Hz | 0.239 (0.263) | 1.133 (0.521)

6. Primary Outcome: End Acceleration Measured in Tibialis Anterior
Description: as for outcome 5
Time Frame: Day 1
Population: 1 subject data set on the No ICU Acquired Weakness Group, could not be analyzed due to excessive subject motion during the trial. One additional subject had no data due to a malfunction with the accelerometer firmware The device manufacturer was contacted and were able to update the device, but no data was recorded during that trial.
Measure: Mean (Standard Deviation); unit: Units of Gravity
Arm/Group | ICU Acquired Weakness Group | No ICU Acquired Weakness Group
Number analyzed (Participants) | 5 | 14
Units of Gravity
  Twitch acceleration at 20 Hz | 0.057 (0.081) | 1.088 (0.703)
  Twitch acceleration at 40 Hz | 0.042 (0.067) | 0.767 (0.517)
  Twitch acceleration at 60 Hz | 0.059 (0.083) | 0.640 (0.565)

7. Primary Outcome: Fatigue Ratio Measured in Extensor Carpi Radialis Longus
Description: Fatigue ratio is the ending acceleration divided by peak acceleration during a given stimulation period. A reference range has not yet been established for this measurement. A higher ratio indicates less change from maximum. A lower score would indicate worse outcome.
Time Frame: Day 1
Population: The team was unable to calculate change for 2 subjects in the ICU Acquired Weakness group. These had palpable contractions, but not large enough to displace the skin above the muscle. 1 subject's results were accidentally deleted and the device manufacturer deemed them unrecoverable. Another subject had no data due to software malfunction, the device manufacturer was able to update the device, but no data was recorded during that trial.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ICU Acquired Weakness Group | No ICU Acquired Weakness Group
Number analyzed (Participants) | 3 | 13
ratio
  Twitch acceleration at 20 Hz | 0.578 (0.266) | 0.862 (0.284)
  Twitch acceleration at 40 Hz | 0.306 (0.194) | 0.562 (0.349)
  Twitch acceleration at 60 Hz | 0.639 (0.136) | 0.707 (0.223)

8. Primary Outcome: Fatigue Ratio Measured in Tibialis Anterior
Description: Fatigue ratio is the ending acceleration divided by peak acceleration during a given stimulation period. A reference range has not yet been established for this measurement.
Time Frame: Day 1
Population: The team was unable to calculate change for 3 subjects in the ICU Acquired Weakness group. These had palpable contractions, but not large enough to displace the skin above the muscle. 1 subject's results were accidentally deleted and the device manufacturer deemed them unrecoverable. Another subject had no data due to software malfunction, the device manufacturer was able to update the device, but no data was recorded during that trial.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ICU Acquired Weakness Group | No ICU Acquired Weakness Group
Number analyzed (Participants) | 2 | 14
ratio
  Twitch acceleration at 2 Hz | 0.610 (0.364) | 0.899 (0.351)
  Twitch acceleration at 4 Hz | 0.471 (0.414) | 0.572 (0.247)
  Twitch acceleration at 6 Hz | 0.437 (0.414) | 0.549 (0.265)

ADVERSE EVENTS:
Time Frame: Day 1
Arm/Group | ICU Acquired Weakness Group | No ICU Acquired Weakness Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/17
Other Adverse Events (participants affected / at risk) | 0/5 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT04166630/Prot_SAP_000.pdf